CLINICAL TRIAL: NCT06829225
Title: A Phase 1, Double-Blind, Placebo-Controlled, Single-Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of MK-7240 in Healthy Chinese Participants.
Brief Title: Single Dose Study of Tulisokibart (MK-7240) in Healthy Chinese Participants (MK-7240-002)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 7240-002; MK-7240-002 (Other: MSD)
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Tulisokibart Dose 1 Treatment Subcutaneous (SC) Injection (Experimental): Participants will receive a single SC injection dose of tulisokibart at dose 1 on Day 1.
  Interventions: Drug: Tulisokibart
- Placebo SC Injection (Placebo Comparator): Participants will receive a single SC injection dose of placebo at on Day 1.
  Interventions: Drug: Placebo
- Tulisokibart Dose 1 Intravenous (IV) Infusion (Experimental): Participants will receive a single IV infusion dose of tulisokibart at dose 1 on Day 1.
  Interventions: Drug: Tulisokibart
- Tulisokibart Dose 2 IV Infusion (Experimental): Participants will receive a single IV infusion dose of tulisokibart at dose 2 on Day 1.
  Interventions: Drug: Tulisokibart
- Tulisokibart Dose 3 IV Infusion (Experimental): Participants will receive a single IV infusion dose of tulisokibart at dose 3 on Day 1.
  Interventions: Drug: Tulisokibart
- Placebo IV Infusion (Placebo Comparator): Participants will receive a single IV infusion dose of placebo on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tulisokibart — SC Injection or IV Infusion
  Other Names: MK-7240
  Arms: Tulisokibart Dose 1 Intravenous (IV) Infusion; Tulisokibart Dose 1 Treatment Subcutaneous (SC) Injection; Tulisokibart Dose 2 IV Infusion; Tulisokibart Dose 3 IV Infusion
Drug: Placebo — Tulisokibart-matched Placebo SC Injection or IV Infusion
  Arms: Placebo IV Infusion; Placebo SC Injection

SUMMARY:
The goal of this study is to learn about the safety of tulisokibart in healthy participants and what happens to tulisokibart over time when participants receive treatment intravenously versus subcutaneously.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria include, but are not limited to:

* Be in good health
* Has a body mass index (BMI) ≥18 and ≤28 kg/m^2 and weight ≥40.0 kg
* Continuous non-smoker who has not used tobacco or nicotine-containing products for at least 3 months prior to the dosing of study drug

Exclusion Criteria:

Exclusion Criteria include, but are not limited to:

* History of cancer (malignancy)
* Has positive serum test for human immunodeficiency virus (HIV), hepatitis C or hepatitis B virus infection

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2024-06-13 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to 99 Days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of the study intervention, whether or not considered related to the study intervention.
Number of Participants Who Discontinued the Study Due to AEs | Up to 99 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of the study intervention, whether or not considered related to the study intervention.
Area Under the Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUC0-last) of Tulisokibart | Predose and at designated timepoints (up to 99 days postdose)
  Blood samples will be collected to determine the AUC0-last of tulisokibart.
Area Under the Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of Tulisokibart | Predose and at designated timepoints (up to 99 days postdose)
  Blood samples will be collected to determine the AUC0-inf of tulisokibart.
Maximum Concentration (Cmax) of Tulisokibart | Predose and at designated timepoints (up to 99 days postdose)
  Blood samples will be collected to determine the Cmax of tulisokibart.
Time to Maximum Concentration (Tmax) of Tulisokibart | Predose and at designated timepoints (up to 99 days postdose)
  Blood samples will be collected to determine the Tmax of tulisokibart.
Apparent Terminal Half-life (t1/2) of Tulisokibart | Predose and at designated timepoints (up to 99 days postdose)
  Blood samples will be collected to determine the t1/2 of tulisokibart.
Apparent Clearance (CL/F) of Tulisokibart | Predose and at designated timepoints (up to 99 days postdose)
  Blood samples will be collected to determine the CL/F of tulisokibart.
Apparent Volume of Distribution (Vz/F) of Tulisokibart | Predose and at designated timepoints (up to 99 days postdose)
  Blood samples will be collected to determine the Vz/F of tulisokibart.

SECONDARY OUTCOMES:
Absolute Bioavailability Expressed as a Percentage (F%) of SC Tulisokibart | Predose and at designated timepoints (up to 99 days postdose)
  Blood samples will be collected to determine the F% of tulisokibart.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Peking University Third Hospital (Site 0001), Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com